CLINICAL TRIAL: NCT03143491
Title: Phase 2a Dose-Rising, Safety, Tolerability, and Efficacy Study of Topical SOR007 for Cervical Intraepithelial Neoplasia (CIN)
Brief Title: Study of SOR007 Ointment for Cervical Intraepithelial Neoplasia (CIN)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study never initiated
Sponsor: DFB Soria, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SOR007-2017-02
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Cervical Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Ointments

STUDY DESIGN:
Intervention Model Description: Phase 2, open-label, dose-rising trial. Subjects will enroll in three dose-rising cohorts of three subjects each. he next dose level cohort will enroll upon a finding of safety and tolerability at the previous cohort's first safety review. If a safety or tolerability issue arises in the first three subjects of a cohort, an additional three subjects will be enrolled at the same dose level. If ≥ 1 of the same safety and tolerability issue recurs in the additional 3 subjects, the prior dose-level will be determined to be the highest dose with an acceptable safety and tolerability profile. If no further safety and tolerability issues are identified in the expanded cohort, dose-escalation will continue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SOR007 0.15% (Experimental): 1 mL of 0.15% SOR007 Ointment
  Interventions: Drug: SOR007 (Uncoated Nanoparticulate Paclitaxel) Ointment
- SOR007 1.0% (Experimental): 1 mL of 1.0% SOR007 Ointment
  Interventions: Drug: SOR007 (Uncoated Nanoparticulate Paclitaxel) Ointment
- SOR007 2.0% (Experimental): 1 mL of 2.0% SOR007 Ointment
  Interventions: Drug: SOR007 (Uncoated Nanoparticulate Paclitaxel) Ointment

INTERVENTIONS:
Drug: SOR007 (Uncoated Nanoparticulate Paclitaxel) Ointment — 1 mL of SOR007 applied topically to the ectocervix once-weekly for four weeks.

SUMMARY:
This is a Phase 2, open-label, dose-rising study evaluating the safety, tolerability, and preliminary efficacy of three concentrations of SOR007 ointment (0.15%, 1.0%, and 2.0%) applied topically once per week for four weeks to the ectocervix of subjects with high grade cervical intraepithelial neoplasia (CIN).

DETAILED DESCRIPTION:
In this Phase 2, open-label, dose-rising study, subjects with high grade (CIN 2 or 3) CIN will receive once-weekly topical application of SOR007 ointment to the ectocervix for four weeks. Subjects will be enrolled in three dose-escalating cohorts of three subjects assigned consecutively to receive 0.15%, 1.0%, or 2.0% SOR007 ointment. At the final study visit (Visit 7) subjects will undergo an excision or punch biopsy to record the stage of CIN. PK samples will be obtained post-application on Day 0 at 1, 2, 4, 6, and 24 hours' post-application on Day 1. Additional PK samples will be collected at each visit. Plasma samples for PK analysis on Days 7, 14 and 21 will be collected prior to SOR007 application.

The Medical Monitor will review all available data prior to dose escalation. Dose-escalation of SOR007 will be determined by the Medical Monitor. This will be repeated for each escalated dose until all dose levels have been enrolled or a dose is determined unsafe. Safety will be assessed in an ongoing manner and formal safety reviews will be conducted twice for each cohort: after Day 14 and after Day 49 of the last subject in the cohort. If a safety or tolerability issue becomes apparent in a cohort, an additional three subjects will be enrolled at that dose level, for a maximum of six subjects in that cohort. If ≥ 1 safety or tolerability issue occurs in the additional 3 subjects, the prior dose-level will be determined to be the highest dose with an acceptable safety and tolerability profile. If no further safety and tolerability issues are identified in the expanded cohort, dose-escalation will continue.

Once the highest dose with an acceptable safety and tolerability profile has been determined by the Medical Monitor, PI, and Sponsor Medical Director, a further 3 subjects will be enrolled to that dose level in order to increase the subject numbers.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent;
* Female adults ≥ 18 years of age;
* Presence of newly diagnosed (within 8 weeks prior to administration of SOR007), histologically confirmed CIN 2, CIN 2/3 or CIN 3;
* Candidate for observation, treatment, or removal of CIN;
* Satisfactory colposcopy (visualization of the entire squamocolumnar junction and margins of any visible lesions);
* Appropriate contraception throughout study period;

Exclusion Criteria:

* Pap smear and/or colposcopy suspicious for invasive disease;
* History of previous conization/LEEP;
* History of toxic shock syndrome;
* Known allergy or prior intolerance to paclitaxel;
* Immunodeficiency (including HIV/AIDS and immunosuppressive medication);
* Current, reported participation in another experimental, interventional protocol;
* Active lower genital infection(s);
* Malignant disease at the time of inclusion, with the exclusion of basal cell carcinoma (BCC) or dermal carcinoma-in-situ;
* Concurrent treatment with cytotoxic, radiation, immune-stimulative, or immune-suppressive therapy, or with systemic corticosteroid dose of > 5 mg/d or prednisone (or its equivalent);
* Concomitant use of topical vaginal medications or products;
* Pregnant or lactating;
* Pregnancy planned within six (6) months following study drug application;
* Significant acute or chronic medical or psychiatric illness or other environmental or social factors that, in the opinion of the Investigator, could compromise subject safety, limit the subject's ability to complete the study, and/or compromise the objectives of the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2017-10-01 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2019-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events | 49 days
  Treatment emergent adverse events will include all reported adverse events, laboratory assessments, physical examination findings, and vital signs.

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the plasma concentration versus time curve (AUC) of SOR007 | 49 days
  Plasma samples for pharmacokinetic (PK) analysis will be obtained on Day 0 at 1, 2, 4, and 6 hours post-application, at 24 hours' post-application (Day 1), and at each subsequent clinic visit (samples on Days 7, 14, and 21 will be obtained prior to dose application).
Pharmacokinetics: Peak plasma concentration (Cmax) of SOR007 | 49 days
  Plasma samples for pharmacokinetic (PK) analysis will be obtained on Day 0 at 1, 2, 4, and 6 hours post-application, at 24 hours' post-application (Day 1), and at each subsequent clinic visit (samples on Days 7, 14, and 21 will be obtained prior to dose application).
Pharmacokinetics: Time at which peak plasma concentration is observed (Tmax) of SOR007 | 49 days
  Plasma samples for pharmacokinetic (PK) analysis will be obtained on Day 0 at 1, 2, 4, and 6 hours post-application, at 24 hours' post-application (Day 1), and at each subsequent clinic visit (samples on Days 7, 14, and 21 will be obtained prior to dose application).
Regression of CIN | Baseline and 49 days
  Colposcopic changes as defined by the modified Reid Colposcopic Index (RCI) and confirmed by biopsy histology

CONTACTS AND LOCATIONS:
Overall Officials: Karen K McCune, MD, PhD, Principal Investigator — University of California, San Francisco; Lisa Rahangdale, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill

IPD SHARING:
Plan to Share IPD: No